CLINICAL TRIAL: NCT05851040
Title: Observation of Wheatgrass and Tulsi Formulation or Its Effect With Allopathic Drugs
Brief Title: Observe the Effect of Wheatgrass and Tulsi Formulation or Individuals Taken With Other Allopathic Drugs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Swalife Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: swalife001
Record Dates: First submitted 2023-04-25; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Blood Pressure, High; Blood Sugar; High; Weight, Birth; Smoking
MeSH Terms: conditions — Hypertension; Hyperglycemia; Birth Weight; Smoking | interventions — Observational Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- With Wheatgrass, tulsi formulation: People using Wheatgrass and Tulsi formulation or individual
  Interventions: Other: Observation study
- With Wheatgrass, tulsi formulation and allopathic drugs: People using Wheatgrass and Tulsi formulations or individuals with chronic disease medicine.
  Interventions: Other: Observation study
- Same age group not using any medication
  Interventions: Other: Observation study

INTERVENTIONS:
Other: Observation study — Looking to find the role of wheatgrass and tulsi give separately or with allopathic drug

SUMMARY:
Antioxidant qualities have been attributed to wheatgrass and tulsi formulation. Free radicals are unstable molecules created by the body during metabolism and exposure to environmental pollutants. Antioxidants are chemicals that can help stop or reduce cell damage caused by these unstable molecules. Oxidative stress, which is brought on by free radicals, has been connected to a number of health issues, including chronic inflammation, cardiovascular disease, cancer, and ageing. Wheatgrass is a rich source of vitamins, minerals, amino acids, and chlorophyll, which have been shown to have antioxidant and anti-inflammatory effects. Tulsi, also known as holy basil, is an herb that has been used in Ayurvedic medicine for centuries and has been found to have antioxidant, anti-inflammatory, and immunomodulatory properties. Several studies have investigated the antioxidant properties of wheatgrass and tulsi formulation. For instance, a study published in the Journal of Food Science and Technology in 2015 found that wheatgrass extract had significant antioxidant activity, as measured by its ability to scavenge free radicals and reduce lipid peroxidation in vitro.

DETAILED DESCRIPTION:
Similarly, a study published in the Journal of Ethnopharmacology in 2001 found that tulsi extract had significant antioxidant activity, as measured by its ability to scavenge free radicals and inhibit lipid peroxidation in vitro. Moreover, a study published in the Journal of Medicinal Food in 2011 investigated the antioxidant and anti-inflammatory effects of a combination of wheatgrass and tulsi extracts in rats. The study found that the combination of wheatgrass and tulsi extracts had significant antioxidant and anti-inflammatory effects, as measured by reductions in oxidative stress markers and pro-inflammatory cytokines. Overall, the available evidence suggests that wheatgrass and tulsi formulations may have antioxidant properties, which could potentially help prevent or slow down oxidative stress-related health problems. However, more research is needed to confirm these findings and determine the optimal dosage and duration of wheatgrass and tulsi formulation use for maximum antioxidant benefits. There are several studies that suggest wheatgrass and tulsi formulations have antioxidant properties. A study evaluated the immunomodulatory and antioxidant properties of a traditional formulation containing Tulsi, ginger, and wheatgrass. Another study investigated the antioxidant potential of anthocyanin extracts from colored wheat flour and wheat-grass juice. Additionally, a synergistic effect of conventional medicinal herbs against oxidative stress was observed in another study that included tulsi and wheatgrass. While a study compared the chemical composition, sensory, phenolic, and antioxidant properties of juices from different wheatgrass and turfgrass species, it did not specifically investigate a formulation with tulsi. Another study found that vitamin C is present in wheatgrass which is also an antioxidant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are having a chronic disease and taking formulation wheat grass and tulsi.
2. Patients who are taking wheatgrass and tulsi separately.
3. Patients who are taking wheatgrass, tulsi and regular medicine. -

Exclusion Criteria:

1. Patients below 30 years.
2. Patients who are having a chronic disease but not using formulations of wheatgrass and tulsi.
3. Patients who are not taking wheatgrass and tulsi separately.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of age group 30 to 65 is targeted who have chronic disease and are taking wheat grass and tulsi formulation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Effect of wheat grass and tulsi in combination on blood pressure | Every four week till 6 months
  Blood Pressure measured in mmHg every four week.
Effect of wheat grass and tulsi in combination on blood sugar | Every four week till 6 months
  Blood Sugar measured in mmol/L every four week
Effect of wheat grass and tulsi in combination on weight | Every four week till 6 months
  Weight is measure in Kg every four week.
Effect of wheat grass and tulsi in combination on smoking | Every four week till 6 months
  questionnaire assesment for "Smoking habits"

SECONDARY OUTCOMES:
Effect of wheat grass and tulsi separately on blood pressure | Every four week till 6 months
  Blood Pressure measured in mmHg every four week.
Effect of wheat grass and tulsi separately on blood sugar | Every four week till 6 months
  Blood Sugar measured in mmol/L every four week.
Effect of wheat grass and tulsi separately on weight | Every four week till 6 months
  Weight is measure in Kg every four week.
Effect of wheat grass and tulsi separately on smoking | Every four week till 6 months
  questionnaire assesment for "Smoking habits"
Effect of wheat grass, tulsi and allopathic drug on blood pressure | Every four week till 6 months
  Blood Pressure measured in mmHg every four week.
Effect of wheat grass, tulsi and allopathic drug on blood sugar | Every four week till 6 months
  Blood Sugar measured in mmol/L every four week.
Effect of wheat grass, tulsi and allopathic drug on weight | Every four week till 6 months
  Weight is measure in Kg every four week.
Effect of wheat grass, tulsi and allopathic drug on smoking | Every four week till 6 months
  questionnaire assesment for "Smoking habits"

CONTACTS AND LOCATIONS:
Locations (1):
- Sinhgad college of Pharmacy, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
We will be sharing the Protocol of the study and the execution.